CLINICAL TRIAL: NCT00600379
Title: A Randomized Controlled Trial of a Virtual Reality Training Program for Ambulatory Patients With Mild-to-moderate Chronic Gait Deficits After Stroke
Brief Title: Virtual Reality Training Program for Ambulatory Patients With Chronic Gait Deficits After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. David Tanne/Director, Stroke Center, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-07-4780-DT-CTIL
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Stroke
Keywords: stroke chronic gait deficits virtual reality training
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A, (Experimental): Virtual Reality training for an overall of 18 sessions 2/week + usual care.
  Interventions: Device: Virtual reality system (CAREN™ Integrated Reality System; MOTEK BV, Netherlands).
- B, (No Intervention): Usual care

INTERVENTIONS:
Device: Virtual reality system (CAREN™ Integrated Reality System; MOTEK BV, Netherlands). — Training 2/w for 9 weeks (total 18 sessions).
  Arms: A,

SUMMARY:
The purpose of this study is to examine the feasibility and efficacy of a virtual reality program for ambulatory patients with mild-to-moderate chronic gait deficits after stroke.

DETAILED DESCRIPTION:
Virtual reality (VR) systems enable the learning of simple and complex skills in a controlled virtual environment; i.e., one in which the different components (constraints) of the environment can be displayed, graded, changed and monitored in a quantitative manner.

Small preliminary studies suggest that VR may be used to augment chronic stroke rehabilitation and may enhance cortical reorganization. Our aim is to examine the feasibility and efficacy of a virtual reality program for ambulatory patients with mild-to-moderate chronic gait deficits after stroke. Study design-a single center randomized controlled trial of an experimental group and a usual care group.

ELIGIBILITY:
Main Inclusion Criteria:

* Stroke within 3-72 months.
* Mild-to-moderate residual gait deficits after the index stroke with preserved capacity for ambulation without or with an assistive device (e.g., walker, cane) or orthotics (e.g. AFO).

Main exclusion Criteria:

* Unstable cardiac or other medical condition or aphasia, dementia or other significant neurological disease limiting ability to train.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Community ambulation using Step Activity Monitor (SAM) | Baseline X2, post training (week 9-10), retention (week 20-24)
Gait analysis (GaitRite system) including dual task | Baseline X2, post training (week 9-10), retention (week 20-24)
Body sway- displacement of center of pressure (CoP) as indicated by the reactive forces from platform. | Baseline X2, post training (week 9-10), retention (week 20-24)
Timed Up and Go | Baseline X2, post training (week 9-10), retention (week 20-24)

SECONDARY OUTCOMES:
Functional Reach | Baseline X2, post training (week 9-10), retention (week 20-24)
Four Stick Stepping Test (FSST) | Baseline X2, post training (week 9-10), retention (week 20-24)
3DGait Analysis system | Baseline X2, post training (week 9-10), retention (week 20-24)
6 minute walk | Baseline X2, post training (week 9-10), retention (week 20-24)
Self-induced perturbations and reaction to perturbations on platform | Baseline X2, post training (week 9-10), retention (week 20-24)

CONTACTS AND LOCATIONS:
Overall Officials: David Tanne, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Strok Center, Tel Litwinsky, Ramat Gan, Israel